CLINICAL TRIAL: NCT06234592
Title: The Effect of Vasopressor Therapy on Renal Perfusion in Patients With Septic Shock - a Mechanistically Focussed Randomized Control Study
Brief Title: The Effect of Vasopressor Therapy on Renal Perfusion in Septic Shock
Acronym: REPERFUSE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: European Society of Intensive Care Medicine (Other); Royal Centre for Defence Medicine (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 328797
Record Dates: First submitted 2024-01-03; First posted 2024-01-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Septic Shock; Acute Kidney Injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury | interventions — Angiotensin II; Vasopressins; Norepinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Angiotensin II Infusion (Experimental): Angiotensin II infusion commenced alongside standard care vasopressor therapy (norepinephrine). Angiotensin II up titrated in a protocolised manner to a target/maximum dose of 40 ng/kg/min whilst noradrenaline down titrated in order to achieve/maintain target mean arterial pressure (MAP) as directed by attending clinician.
  Interventions: Drug: Angiotensin II; Drug: Norepinephrine
- Vasopressin Infusion (Experimental): Vasopressin infusion commenced alongside standard care vasopressor therapy (norepinephrine). Vasopressin up titrated in a protocolised manner to a target/maximum dose of 0.04 IU/min whilst noradrenaline down titrated in order to achieve/maintain target mean arterial pressure (MAP) as directed by attending clinician.
  Interventions: Drug: Vasopressin; Drug: Norepinephrine
- Norepinephrine Infusion (Active Comparator): Standard care vasopressor therapy which recruited participants already receiving, titrated to achieve/maintain target mean arterial pressure (MAP) as directed by attending clinician.
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Angiotensin II — Angiotensin II infusion
  Arms: Angiotensin II Infusion
Drug: Vasopressin — Vasopressin infusion
  Arms: Vasopressin Infusion
Drug: Norepinephrine — Standard care vasopressor therapy, norepinephrine infusion

SUMMARY:
Acute kidney injury (AKI) is a common complication of septic shock and together these conditions carry a high mortality risk. In septic patients who develop severe AKI renal cortical perfusion is deficient despite normal macrovascular organ blood flow. This intra-renal perfusion abnormality may be amenable to pharmacological manipulation, which may offer mechanistic insight into the pathophysiology of septic AKI. The aim of the current study is to investigate the effects of vasopressin and angiotensin II on renal microcirculatory perfusion in a cohort of patients with septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Within 48 hours of intensive care admission
* Evidence of suspected or confirmed infection
* Sequential Organ Failure (SOFA) score increase of 2 or more (assuming a baseline of 0 if no previous measures)
* Requirement for norepinephrine infusion as the sole vasopressor agent in a dose of >0.1mcg/kg/min
* Lactate >2mmol/L at any stage prior to randomisation

Exclusion Criteria:

* Known intolerance to Sonovue™ contrast medium, vasopressin or angiotensin II
* Patients receiving other vasoactive drugs in addition to norepinephrine
* Patients with known chronic kidney disease (CKD) stage 4 or 5 (baseline glomerular filtration rate (GFR) <30mls/min)
* Patients receiving extra corporal membrane oxygenation (ECMO)
* Patients with acute occlusive coronary syndromes requiring intervention
* Patients with mesenteric ischaemia
* Patients with a history or presence of aortic dissection or abdominal aortic aneurysm
* Patients with Raynaud's syndrome or acute vaso-occlusive conditions
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-01-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Cortical mean transit time (mTT) measured in seconds | Measured at +24 hours following study vasopressor infusion starting
  Contrast enhanced ultrasound measure of renal cortical tissue blood flow

SECONDARY OUTCOMES:
Cortical mean transit time (mTT) measured in seconds | Measured at +1 hour and +24 hours following study vasopressor infusion starting
  Contrast enhanced ultrasound measures of renal cortical tissue blood flow
Cortical perfusion index (PI) measured in arbitrary units | Measured at +1 hour and +24 hours following study vasopressor infusion starting
  Contrast enhanced ultrasound measures of renal cortical tissue blood flow
Cortical wash in rate (WiR) measured in arbitrary units | Measured at +1 hour and +24 hours following study vasopressor infusion starting
  Contrast enhanced ultrasound measures of renal cortical tissue blood flow
Urinary oxygen tension (pO2) across 24 hours study period measured in millimetres of mercury (mmHg) | Across 24 hours study period
  Mean urinary pO2
Tissue inhibitor of metalloproteinases-2 (TIMP-2) and insulin-like growth factor binding protein-7 (IGFBP-7). Both measured in nanograms per millilitre (ng/ml) | Measured at baseline and +24 hours following study vasopressor infusion starting
  Biomarker analysis - regulatory proteins involved in initiating cell cycle arrest and associated with AKI

OTHER OUTCOMES:
Perfused vessel density (PVD) measured in millimetres per square millimetre | Measured at +1 hour and +24 hours following study vasopressor infusion starting
  Incident dark field video microscopy measures of the systemic microcirculation
Microvascular flow index (MFI) (unitless score from 0 to 3 where 3 is the value see in health). | Measured at +1 hour and +24 hours following study vasopressor infusion starting
  Incident dark field video microscopy measures of the systemic microcirculation
Syndecan 1, angiopoietin 1 & 2, Interleukin 6 & 8 (IL-6, IL-8) and tissue necrosis factor (TNF). All measured in nanograms per millilitre (ng/ml) | Measured at baseline and +24 hours following study vasopressor infusion starting
  Biomarker analysis - markers of inflammation and endothelial activation/function

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] McDonald R, Watchorn J, Mehta R, Ostermann M, Hutchings S. The REPERFUSE study protocol: The effects of vasopressor therapy on renal perfusion in patients with septic shock-A mechanistically focused randomised control trial. PLoS One. 2024 Jun 13;19(6):e0304227. doi: 10.1371/journal.pone.0304227. eCollection 2024. PMID 38870103